CLINICAL TRIAL: NCT02450578
Title: Evaluation of the Prophylactic Antimalarial Activity of a Single Dose of DSM265 in Non-immune Healthy Adult Volunteers by Controlled Human Malaria Infection With PfSPZ Challenge
Brief Title: DSM265 Chemoprophylaxis of Plasmodium Falciparum Malaria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Institute of Tropical Medicine, University of Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MMV_DSM265_14_01
Record Dates: First submitted 2015-03-16; First posted 2015-05-21 (Estimated); Results first posted 2020-12-03 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Plasmodium Falciparum, Malaria
Keywords: Malaria, Plasmodium falciparum sporozoite challenge, DSM265
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — DSM265; atovaquone, proguanil drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1a: DSM265/placebo, sporozoite inoculum (Experimental): DSM265 400mg / placebo Day -1, sporozoite inoculum Day 0
  Interventions: Drug: DSM265 400mg; Drug: Placebo to DSM265 400 mg; Biological: Plasmodium falciparum sporozoite challenge
- Cohort 1b: Malarone, sporozoite inoculum (Active Comparator): Malarone daily for 9 days from Day -1 to Day 7, sporozoite inoculum Day 0
  Interventions: Biological: Plasmodium falciparum sporozoite challenge; Drug: Malarone
- Cohort 2: DSM265/placebo, sporozoite inoculum (Experimental): DSM265 400mg / placebo Day -7, sporozoite inoculum Day 0
  Interventions: Drug: DSM265 400mg; Drug: Placebo to DSM265 400 mg; Biological: Plasmodium falciparum sporozoite challenge
- Cohort 3: DSM265 / placebo, sporozoite inoculum (Optional) (Experimental): DSM265 400mg / placebo Day -X, sporozoite inoculum Day 0
  Interventions: Drug: DSM265 400mg; Drug: Placebo to DSM265 400 mg; Biological: Plasmodium falciparum sporozoite challenge

INTERVENTIONS:
Drug: DSM265 400mg — DSM265 400mg, single oral administration in a fed state
  Arms: Cohort 1a: DSM265/placebo, sporozoite inoculum; Cohort 2: DSM265/placebo, sporozoite inoculum; Cohort 3: DSM265 / placebo, sporozoite inoculum (Optional)
Drug: Placebo to DSM265 400 mg — Placebo to DSM265 400mg, single oral administration in a fed state
  Arms: Cohort 1a: DSM265/placebo, sporozoite inoculum; Cohort 2: DSM265/placebo, sporozoite inoculum; Cohort 3: DSM265 / placebo, sporozoite inoculum (Optional)
Biological: Plasmodium falciparum sporozoite challenge — IV Plasmodium falciparum sporozoites (3200) by direct venous inoculation
  Other Names: Sporozoite inoculum
Drug: Malarone — 250 mg atovaquone, 100 mg proguanil hydrochloride
  Other Names: atovaquone / proguanil hydrochloride
  Arms: Cohort 1b: Malarone, sporozoite inoculum

SUMMARY:
Study to evaluate the efficacy of DSM265 as a causal prophylactic in a standardized and validated Human Challenge model using direct venous inoculation of aseptic, purified, cryopreserved, vialed Plasmodium falciparum sporozoites.

DETAILED DESCRIPTION:
This study follows the First In Human dose-escalation study of DSM265 (25 - 800 mg of DSM265) and an Induced-Blood Stage Malaria Challenge study (150 mg of DSM265) conducted in healthy adult volunteers in Australia. After identification of efficacious DSM265 plasma concentrations in the Induced-Blood Stage Malaria model, the current study will evaluate the efficacy of DSM265 as a causal prophylactic in a standardized and validated Human Challenge model using direct venous inoculation of aseptic, purified, cryopreserved, vialed Plasmodium falciparum sporozoites (Challenge).

Three sequential cohorts of healthy male and women volunteers, of non-childbearing potential or of childbearing potential with predefined accepted methods of contraception, are planned in order to investigate three preventive conditions with regard to administration of DSM265. Preventive administration of the study drug will occur 1 and 7 days before inoculum of Plasmodium falciparum sporozoite Challenge, with a last cohort administered at a time point to be determined from the 2 previous cohorts but which will not exceed 28 days before the challenge. The study will also include a cohort where subjects will be treated with atovaquone-proguanil (Malarone®) using the approved regimen for chemoprophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Good health based on medical history and physical examination- Body mass index >18 and <30 kg/m2
* Lab results without clinically significant findings in 28 days prior to enrolment
* Negative drug screening test
* Females: negative pregnancy test at screening and on the day before first dose of DSM265 and sporozoite challenge injection
* Sexually active males must agree to use a medically acceptable form of contraception from enrolment and continue for 12 weeks after the dose of DSM265
* Women may only be included if they are either Identified as not of child bearing potential, or if of child bearing potential and willing and able to practice one of the continuous acceptable methods of contraception (must be one with failure rate less than 1% per year) with double barrier protection:

  * Intrauterine device+condoms,
  * Diaphragms+spermicidal gel/foam+condoms,
  * Hormonal contraceptives (oral, depot, patch, injectable or vaginal ring) stabilized for at least 30 days before the study drug + condoms from screening to at least 60 days after dose of DSM265
* Agree to allow the investigators to discuss the medical history with General Practitioner and to sign a request to release medical information concerning contra-indications for participation in the study
* Able and willing to comply with all study requirements for the duration of the study
* Agree to undergo all study procedures, to attend all study visits and stay overnight for observation if required, up to last follow up visit
* Willing to undergo a sporozoite challenge
* Able and willing to answer all questions on the informed consent quiz correctly demonstrating an understanding of the meaning and of the study procedures
* Able and willing to sign the informed consent form
* Reachable (24/7) by mobile phone or email during the whole study period
* Agree to refrain from blood donation during the course of the study and after the end of involvement in the study according to the local and national blood banking eligibility criteria (currently 4 years in Germany)
* Willing to take a curative regimen of Riamet or another registered antimalarial if necessary

Exclusion Criteria:

* Any history of malaria
* Plans to travel to malaria endemic region during the study period up to last follow up visit or plans to travel outside of Germany during the challenge period
* unable to be closely followed for social, geographic or psychological reasons
* Previous participation in any malaria vaccine study or controlled human malaria infection study
* Participation in any other clinical study within 30 days before enrolment in the study, or plan to participate in another investigational vaccine/drug research during the study period.
* Woman who is breast-feeding or planning to become pregnant during the study
* Positive human immunodeficiency virus, seropositive for hepatitis B surface antigen or Hepatitis C virus tests
* Any confirmed/suspected immunosuppressive or immunodeficient state, including human immunodeficiency virus infection, asplenia, recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the 6 months before enrolment (inhaled and topical steroids are allowed)
* History of serious psychiatric condition that may affect participation in the study, precludes compliance with the protocol; past or present psychoses; disorder requiring lithium; or within 5 years prior to enrolment, history of a suicide plan or attempt.
* History of convulsions or severe head trauma
* Symptoms, physical signs and lab values suggestive of systemic disorders including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, and other conditions which could interfere with the interpretation of the study results or compromise health
* History of cancer (except basal cell carcinoma of the skin), or diabetes mellitus or of arrhythmias or documented prolonged QTF-interval (>450msec)
* Clinically significant abnormalities in electrocardiogram at screening: pathologic Q wave, prolonged QT interval, and significant ST-T wave changes, left ventricular hypertrophy, non-sinus rhythm except isolated premature atrial contractions, right or left bundle branch block, advanced A-V heart block (type 2 or type 3)
* In moderate risk or higher categories for fatal or non-fatal cardiovascular event within 5 years (>10%) determined by non-invasive criteria for cardiac risk
* Positive family history in relatives <50 years for cardiac disease
* History of psoriasis or porphyria, which may be exacerbated by chloroquine
* History of splenectomy
* Sickle cell anaemia or other red blood cell disorders
* History of allergy or contra-indications to or having contraindications to the use of chloroquine phosphate, atovaquone-proguanil (cohort 1B), artemether or lumefantrine
* Use of any prescription drugs (except contraception), herbal supplements or over-the-counter medication in 4 weeks before dosing or 5x half-lives, whichever is longer
* Use or anticipated use of medications known to cause drug reactions with rescue medications or Malarone, such as cimetidine, metoclopramide, antacids and taken at any point during the study period.
* Intake of grapefruit, grapefruit juice, Seville orange or other products containing these ingredients within 7 days of the first drug administration
* Use of chronic immunosuppressive drugs, or other immune modifying drugs within 6 months of enrolment (inhaled and topical corticosteroids and oral anti-histaminic are allowed) and/or during the study period
* Use of systemic antibiotics with known antimalarial activity within 30 days of study enrolment (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones, or azithromycin ) and/or during the study period
* Use of immunoglobulins or blood products in 3 months prior to enrolment
* Suspected/known injecting drug abuse in 5 years preceding enrolment
* Current smoking more than 10 cigarettes or equivalent per day
* Plan for major surgery between enrolment and follow up

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Mordmüller, Dr. med, Principal Investigator — Institut für Tropenmedizin, Uni. of Tübingen
Locations (1):
- Universitätsklinikum Tübingen, Institut für Tropenmedizin, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sulyok M, Ruckle T, Roth A, Murbeth RE, Chalon S, Kerr N, Samec SS, Gobeau N, Calle CL, Ibanez J, Sulyok Z, Held J, Gebru T, Granados P, Bruckner S, Nguetse C, Mengue J, Lalremruata A, Sim BKL, Hoffman SL, Mohrle JJ, Kremsner PG, Mordmuller B. DSM265 for Plasmodium falciparum chemoprophylaxis: a randomised, double blinded, phase 1 trial with controlled human malaria infection. Lancet Infect Dis. 2017 Jun;17(6):636-644. doi: 10.1016/S1473-3099(17)30139-1. Epub 2017 Mar 28. PMID 28363637

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 40 subjects were screened. Of these 22 (55.0%) were enrolled to participate in the study
Pre-assignment Details: One subject was allocated to treatment but did not receive any study medication due to an ECG abnormality discovered after randomization and, therefore, 21 out of 22 subjects received at least one dose of the study medications.
  In agreement with the Safety Review Team, the Sponsor decided to close the study without progressing to conduct Cohort 3.
Groups:
- Cohort 1A: 400 mg DSM265, Sporozoite Challenge: DSM265 400mg on Day -1, sporozoite challenge on Day 0
  DSM265 400mg: single oral administration in a fed state
  Plasmodium falciparum sporozoite challenge: Plasmodium falciparum sporozoites (3200) by direct venous inoculation
- Cohort 1B: Malarone, Sporozoite Challenge: Malarone daily for 9 days from Day -1 to Day 7, sporozoite challenge Day 0
  Malarone: 250 mg atovaquone, 100 mg proguanil hydrochloride
  Plasmodium falciparum sporozoite challenge: Plasmodium falciparum sporozoites (3200) by direct venous inoculation
- Cohort 2: 400 mg DSM265, Sporozoite Challenge: DSM265 400mg on Day -7, sporozoite challenge on Day 0
  DSM265 400mg: single oral administration in a fed state
  Plasmodium falciparum sporozoite challenge: Plasmodium falciparum sporozoites (3200) by direct venous inoculation
- Placebo Cohorts 1A and 2, Sporozoite Challenge: Placebo to DSM265 400 mg on Day -1, sporozoite challenge on Day 0
  Placebo: Single oral administration in a fed state
  Plasmodium falciparum sporozoite challenge: Plasmodium falciparum sporozoites (3200) by direct venous inoculation
Period: Overall Study
Arm/Group | Cohort 1A: 400 mg DSM265, Sporozoite Challenge | Cohort 1B: Malarone, Sporozoite Challenge | Cohort 2: 400 mg DSM265, Sporozoite Challenge | Placebo Cohorts 1A and 2, Sporozoite Challenge
Started | 6 | 6 | 6 | 4
Completed | 5 | 6 | 6 | 4
Not Completed | 1 | 0 | 0 | 0
Not completed — ECG abnormality so not treated | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: one subject in cohort 1A was excluded prior to dosing
Groups:
- Cohort 1A: 400 mg DSM265, Sporozoite Challenge: DSM265 400 mg on Day -1, sporozoite challenge on Day 0
  DSM265 400 mg: single oral administration in a fed state
  Plasmodium falciparum sporozoite challenge: Plasmodium falciparum sporozoites (3200) by direct venous inoculation
- Cohort 2: 400 mg DSM265, Sporozoite Challenge: DSM265 400 mg on Day -7, sporozoite challenge on Day 0
  DSM265 400 mg: single oral administration in a fed state
  Plasmodium falciparum sporozoite challenge: Plasmodium falciparum sporozoites (3200) by direct venous inoculation
- Placebo Cohorts 1A and 2: Placebo to DSM265 400 mg on Day -7, sporozoite challenge on Day 0
  Placebo to DSM265 400 mg: single oral administration in a fed state
  Plasmodium falciparum sporozoite challenge: Plasmodium falciparum sporozoites (3200) by direct venous inoculation
- Total: Total of all reporting groups
Arm/Group | Cohort 1A: 400 mg DSM265, Sporozoite Challenge | Cohort 1B: Malarone, Sporozoite Challenge | Cohort 2: 400 mg DSM265, Sporozoite Challenge | Placebo Cohorts 1A and 2 | Total
Number analyzed (Participants) | 5 | 6 | 6 | 4 | 21
Age, Customized [Mean (Standard Deviation); unit: years]
  Age (years) | 24.20 (4.02) | 26.67 (4.93) | 25.33 (4.18) | 24.82 (3.95) | 26.00 (4.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 2 | 8
  Male | 3 | 4 | 4 | 2 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 5 | 6 | 6 | 4 | 21
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 5 | 6 | 6 | 4 | 21

OUTCOME MEASURES:

1. Primary Outcome: Infection Rate
Description: The infection rate is the number (percentage) of subjects in a cohort who became positive for parasitemia.
  Complete protection = Subjects with pre-patent period equal to 28 days.
Time Frame: Day 0 to Day 28 post-inoculum (daily)
Population: All subjects who received both at least one dose of study medication and the PfSPZ challenge
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1A: 400 mg DSM265 (Day-1), Sporozoite Challenge (Day0): DSM265 400 mg on Day -1, sporozoite challenge on Day 0
  DSM265 400 mg: single oral administration in a fed state
  Plasmodium falciparum sporozoite challenge: Plasmodium falciparum sporozoites (3200) by direct venous inoculation
- Cohort 2: 400 mg DSM265 (Day-7), Sporozoite Challenge (Day0): DSM265 400 mg on Day -7, sporozoite challenge on Day 0
  DSM265 400 mg: single oral administration in a fed state
  Plasmodium falciparum sporozoite challenge: Plasmodium falciparum sporozoites (3200) by direct venous inoculation
- Placebo Cohorts 1A and 2: Placebo to DSM265 400 mg on Day -7 or Day -1, sporozoite challenge on Day 0
  Placebo to DSM265 400 mg: single oral administration in a fed state
  Plasmodium falciparum sporozoite challenge: Plasmodium falciparum sporozoites (3200) by direct venous inoculation
Arm/Group | Cohort 1A: 400 mg DSM265 (Day-1), Sporozoite Challenge (Day0) | Cohort 1B: Malarone, Sporozoite Challenge | Cohort 2: 400 mg DSM265 (Day-7), Sporozoite Challenge (Day0) | Placebo Cohorts 1A and 2
Number analyzed (Participants) | 5 | 6 | 6 | 4
Participants
  Complete Protection | 5 | 6 | 3 | 0
  Parasitemic | 0 | 0 | 3 | 4

2. Primary Outcome: Pre-patent Period
Description: The pre-patent period is defined as the time (days) from inoculation with PfSPZ to first occurrence of a positive TBS. If no positive TBS is seen by Day 28, this variable is set to 28 days.
  Complete protection = Subjects showing with pre-patent period equal to 28 days.
Time Frame: Day 0 to Day 28 post-inoculum (daily)
Population: All subjects who received both at least one dose of study medication and the PfSPZ challenge
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | Cohort 1A: 400 mg DSM265 (Day-1), Sporozoite Challenge (Day0) | Cohort 1B: Malarone, Sporozoite Challenge | Cohort 2: 400 mg DSM265 (Day-7), Sporozoite Challenge (Day0) | Placebo Cohorts 1A and 2
Number analyzed (Participants) | 5 | 6 | 6 | 4
Days | 28.0 (0.00) | 28.0 (0.00) | 20.6 (2.78) | 11.7 (7.93)

3. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety & Tolerability of DSM265
Description: Safety & tolerability of DSM265 for causal and suppressive chemoprophylaxis in non-immune healthy volunteers in a non-immune healthy volunteers in CHMI with PfSPZ challenge.
Time Frame: From first dose (Day -1 in Cohort 1A and Day -7 in Cohort 2) to Day 60 post-inoculum
Population: All the subjects included in the safety population were administered the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a: DSM265/Placebo, Sporozoite Inoculum | Cohort 2: DSM265/Placebo, Sporozoite Inoculum
Number analyzed (Participants) | 5 | 6
Participants | 5 | 6

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) as a Measure of Safety & Tolerability of Malarone
Description: Safety & tolerability of Malarone for causal and suppressive chemoprophylaxis in non-immune healthy volunteers in a Plasmodium falciparum sporozoite challenge. Measured by adverse events, laboratory data.
  Malarone® was administered as a single daily dose over a period of 9 days from Day -1 to Day 7.
Time Frame: From first dose (Day -1, Cohort 1b) to Day 60 post-inoculum
Population: All the subjects included in the safety population were administered the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1B: Malarone, Sporozoite Challenge
Number analyzed (Participants) | 6
Participants | 5

5. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability of Plasmodium Falciparum Sporozoite Challenge Inoculum
Description: Safety & tolerability of Plasmodium falciparum sporozoite challenge inoculum during DSM265 administration, and Malarone administration. Measured by adverse events, laboratory data
Time Frame: Day 0 to Day 60 post-inoculum
Population: All the subjects included in the safety population were administered the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A: 400 mg DSM265 (Day-1), Sporozoite Challenge (Day0) | Cohort 1B: Malarone, Sporozoite Challenge | Cohort 2: 400 mg DSM265 (Day-7), Sporozoite Challenge (Day0) | Placebo Cohorts 1A and 2
Number analyzed (Participants) | 5 | 6 | 6 | 4
Participants | 3 | 5 | 5 | 4

6. Secondary Outcome: DSM265 Pharmacokinetics Profile - T Max
Description: Pre-dose and post-dose during the period including Day 28
Time Frame: From pre-dose of DSM265 (Day -1 in Cohort 1a and Day -7 in Cohort 2) to Day 28 post-inoculum
Population: All subjects who received study drug and provided they had sufficient DSM265 and/or DSM450 concentration data for the non-compartmental analysis were included in the pharmacokinetic analysis (all-treated set).
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1A: 400 mg DSM265 (Day-1), Sporozoite Challenge (Day0) | Cohort 2: 400 mg DSM265 (Day-7), Sporozoite Challenge (Day0)
Number analyzed (Participants) | 5 | 6
hours
  T max DBS | 2.02 [1.00 to 14.0] | 8.48 [0.500 to 14.0]
  T max Plasma | 2.00 [1.00 to 4.02] | 8.48 [0.500 to 14.0]

7. Secondary Outcome: DSM265 Pharmacokinetics Profile - T 1/2
Description: Pre-dose and post-dose during the period including Day 28
Time Frame: From pre-dose of DSM265 (Day -1 in Cohort 1a and Day -7 in Cohort 2) to Day 28 post-inoculum
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Cohort 1A: 400 mg DSM265 (Day-1), Sporozoite Challenge (Day0) | Cohort 2: 400 mg DSM265 (Day-7), Sporozoite Challenge (Day0)
Number analyzed (Participants) | 5 | 6
hours
  t 1/2 DBS | 132 (31.4) | 113 (39.0)
  t 1/2 Plasma | 134 (34.8) | 116 (40.4)

8. Secondary Outcome: DSM265 Pharmacokinetics Profile - C Max
Description: Pre-dose and post-dose during the period including Day 28
Time Frame: From pre-dose of DSM265 (Day -1 in Cohort 1a and Day -7 in Cohort 2) to Day 28 post-inoculum
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1A: 400 mg DSM265 (Day-1), Sporozoite Challenge (Day0) | Cohort 2: 400 mg DSM265 (Day-7), Sporozoite Challenge (Day0)
Number analyzed (Participants) | 5 | 6
ng/mL
  C max DBS | 6860 (28.2) | 6990 (15.0)
  C max Plasma | 13300 (34.3) | 11200 (18.0)

9. Secondary Outcome: DSM265 Pharmacokinetics Profile - AUC 0-∞, AUC 0-168h, and AUC 0-480h
Description: Pre-dose and post-dose during the period including Day 28 for AUC 0-∞, AUC 0-168h, and AUC 0-480h
Time Frame: From pre-dose of DSM265 (Day -1 in Cohort 1a and Day -7 in Cohort 2) to Day 28 post-inoculum
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Cohort 1A: 400 mg DSM265 (Day-1), Sporozoite Challenge (Day0) | Cohort 2: 400 mg DSM265 (Day-7), Sporozoite Challenge (Day0)
Number analyzed (Participants) | 5 | 6
ng*h/mL
  AUC 0-∞ DBS | 979000 (25.8) | 906000 (29.8)
  AUC 0-∞ Plasma | 1870000 (23.4) | 1540000 (30.4)
  AUC 0-168h DBS | 582000 (22.8) | 568000 (13.3)
  AUC 0-168h Plasma | 1100000 (22.3) | 949000 (14.0)
  AUC 0-480h DBS | 863000 (22.0) | 847000 (25.4)
  AUC 0-480h Plasma | 1680000 (19.5) | 1430000 (25.9)

10. Secondary Outcome: DSM265 Pharmacokinetics Profile - CL/F
Description: Pre-dose and post-dose during the period including Day 28
Time Frame: From pre-dose of DSM265 (Day -1 in Cohort 1a and Day -7 in Cohort 2) to Day 28 post-inoculum
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | Cohort 1A: 400 mg DSM265 (Day-1), Sporozoite Challenge (Day0) | Cohort 2: 400 mg DSM265 (Day-7), Sporozoite Challenge (Day0)
Number analyzed (Participants) | 5 | 6
mL/h
  CL/F DBS | 409 (25.8) | 441 (29.8)
  CL/F Plasma | 214 (23.4) | 260 (30.4)

11. Secondary Outcome: DSM265 Pharmacokinetics Profile - Vz/F
Description: Pre-dose and post-dose during the period including Day 28
Time Frame: From pre-dose of DSM265 (Day -1 in Cohort 1a and Day -7 in Cohort 2) to Day 28 post-inoculum
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | Cohort 1A: 400 mg DSM265 (Day-1), Sporozoite Challenge (Day0) | Cohort 2: 400 mg DSM265 (Day-7), Sporozoite Challenge (Day0)
Number analyzed (Participants) | 5 | 6
mL
  Vz/F DBS | 77900 (29.0) | 71700 (18.7)
  Vz/F Plasma | 41400 (31.8) | 43600 (18.9)

12. Secondary Outcome: DSM450 Pharmacokinetics Profile - T Max
Description: Pre-dose and post-dose during the period including Day 28
Time Frame: From pre-dose of DSM265 (Day -1 in Cohort 1a and Day -7 in Cohort 2) to Day 28 post-inoculum
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1A: 400 mg DSM265 (Day-1), Sporozoite Challenge (Day0) | Cohort 2: 400 mg DSM265 (Day-7), Sporozoite Challenge (Day0)
Number analyzed (Participants) | 5 | 6
hours
  t max DBS | 169 [71.9 to 265] | 216 [48.3 to 267]
  t max Plasma | 169 [71.9 to 265] | 169 [72.4 to 266]

13. Secondary Outcome: DSM450 Pharmacokinetics Profile - Cmax
Description: Pre-dose and post-dose during the period including Day 28
Time Frame: From pre-dose of DSM265 (Day -1 in Cohort 1a and Day -7 in Cohort 2) to Day 28 post-inoculum
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1A: 400 mg DSM265 (Day-1), Sporozoite Challenge (Day0) | Cohort 2: 400 mg DSM265 (Day-7), Sporozoite Challenge (Day0)
Number analyzed (Participants) | 5 | 6
ng/mL
  Cmax DBS | 545 (35.3) | 714 (37.1)
  Cmax Plasma | 999 (31.0) | 1170 (36.7)

14. Secondary Outcome: DSM450 Pharmacokinetics Profile - AUC 0-t, AUC 0-168h, and AUC 0-480h
Description: Pre-dose and post-dose during the period including Day 28 for AUC 0-t, AUC 0-168h, and AUC 0-480h
Time Frame: From pre-dose of DSM265 (Day -1 in Cohort 1a and Day -7 in Cohort 2) to Day 28 post-inoculum
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Cohort 1A: 400 mg DSM265 (Day-1), Sporozoite Challenge (Day0) | Cohort 2: 400 mg DSM265 (Day-7), Sporozoite Challenge (Day0)
Number analyzed (Participants) | 5 | 6
ng*h/mL
  AUC 0-∞ DBS | 185000 (34.9) | 225000 (42.5)
  AUC 0-∞ Plasma | 326000 (32.1) | 367000 (39.7)
  AUC 0-168h DBS | 63800 (44.9) | 85300 (45.1)
  AUC 0-168h Plasma | 115000 (45.9) | 142000 (40.4)
  AUC 0-480h DBS | 185000 (34.9) | 234000 (46.5)
  AUC 0-480h Plasma | 326000 (32.1) | 375000 (44.1)

15. Secondary Outcome: The Pharmacokinetic-pharmacodynamic Profile of Pre-administration of DSM265 on Clearance of Plasmodium Falciparum Parasites After Administration of the Sporozoite Challenge
Description: The profile of plasma concentrations and pharmacokinetic parameters (AUC, Cmax, Tmax, T0-inf, AUC0-t, t1/2) will be reviewed on a background of the safety profile (adverse events, laboratory and ECG data) and the clearance of Plasmodium falciparum parasites (efficacy) after administration of the sporozoite challenge
Time Frame: From first dose of DSM265 (Day -1 in Cohort 1a, Day -7 in Cohort 2 and Day -X in Cohort 3) to 480 hours post-dose
Population: Data were not collected. Analysis was not done because, because all subjects were administered with the same dose of 400mg DSM; so not enough variability for the "DSM concentration" parameter.
Arm/Group | Cohort 1A: 400 mg DSM265 (Day-1), Sporozoite Challenge (Day0) | Cohort 2: 400 mg DSM265 (Day-7), Sporozoite Challenge (Day0)
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Recrudescence of Parasite Kinetics Following DSM265 Administration.
Description: On any re-appearance of parasites, thick smears and PCR samples will be examined to determine whether the parasite is a different variant(recrudescence) or has the same genetic profile as the original infection (re-infection) post-dose
Time Frame: Day 6 post-inoculum to Day 60
Population: Recrudescence was not observed in this study.
Arm/Group | Cohort 1A: 400 mg DSM265 (Day-1), Sporozoite Challenge (Day0) | Cohort 2: 400 mg DSM265 (Day-7), Sporozoite Challenge (Day0)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the day of dosing until Day 60 following PfSPZ challenge: Cohort 1A: 61 days Cohort 1B (Malarone): 61 days Cohort 2: 68 days
Arm/Group | Cohort 1A: 400 mg DSM265 (Day-1), Sporozoite Challenge (Day0) | Cohort 1B: Malarone, Sporozoite Challenge | Cohort 2: 400 mg DSM265 (Day-7), Sporozoite Challenge (Day0) | Placebo Cohorts 1A and 2
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/6 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 5/5 | 5/6 | 6/6 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1A: 400 mg DSM265 (Day-1), Sporozoite Challenge (Day0) (N=5) | Cohort 1B: Malarone, Sporozoite Challenge (N=6) | Cohort 2: 400 mg DSM265 (Day-7), Sporozoite Challenge (Day0) (N=6) | Placebo Cohorts 1A and 2 (N=4)
Pulmonary embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — One SAE was reported (pulmonary embolism) which was considered to be unrelated to the study drug due to identified risk factors (oral contraception, transatlantic flight) and timing of event (34 days after treatment intake).
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1A: 400 mg DSM265 (Day-1), Sporozoite Challenge (Day0) (N=5) | Cohort 1B: Malarone, Sporozoite Challenge (N=6) | Cohort 2: 400 mg DSM265 (Day-7), Sporozoite Challenge (Day0) (N=6) | Placebo Cohorts 1A and 2 (N=4)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (4)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 4 (5) | 2 (2)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Fatigue (General disorders) | 1 (1) | 1 (1) | 6 (10) | 4 (7)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 3 (8) | 2 (6)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (4) | 2 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Headache (Nervous system disorders) | 1 (2) | 1 (1) | 5 (11) | 4 (11)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No